CLINICAL TRIAL: NCT04875741
Title: Comparative Effects of Neural Mobilization and Muscle Energy Technique on Pain, Range of Motion and Functional Disability in Patients With Sciatica:A Randomized Controlled Trial
Brief Title: Comparative Effects of Neural Mobilization and Muscle Energy Technique in Sciatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/826/2021
Record Dates: First submitted 2021-04-26; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Acute Sciatica; Pain
Keywords: Neural mobilization; Muscle energy technique; Sciatica
MeSH Terms: conditions — Pain; Sciatica

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study would be double-blind as the identity of the patient's group will not be revealed to the assessor and the patient will also be un-aware of the group to which they will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural mobilization (Active Comparator): Patient in this study group will get 30 minutes session, twice weekly for 6 weeks. Neural mobilization technique will be applied to the subjects in addition to conventional treatment.
  Interventions: Other: Neural mobilization
- Muscle energy technique (Experimental): Patient in this study group will get 30 minutes session, twice weekly for 6 weeks. Muscle energy technique will be applied to the subjects in addition to conventional treatment.
  Interventions: Other: Muscle energy technique

INTERVENTIONS:
Other: Neural mobilization — Mobilization of the structures within and around the nervous system is broadly known as Neural Mobilization.
  Other Names: Rehabilitation following Neural Mobilization
  Arms: Neural mobilization
Other: Muscle energy technique — Manual therapy technique initially developed and used by the osteopaths is known as Muscle energy techniques(MET).This technique is effective for the pain reduction, lengthening of the shortened muscle and fascia, improvement in blood circulation and promoting lymph drainage.
  Other Names: Rehabilitation following muscle energy technique
  Arms: Muscle energy technique

SUMMARY:
In this study, investigator will see the effects of neural mobilization in comparison to the muscle energy technique in the patients suffering from sciatica. Impact of the these two interventional techniques , there out come measures i.e pain, range of motion and functional disability.

DETAILED DESCRIPTION:
This study is aimed in comparison among two interventional techniques i.e neural mobilization and muscle energy technique patients with sciatica. This study will be a randomized controlled trial with double blinded protocol, patients will be randomly allocated in to the two groups. one is the neural mobilization technique group and other is the muscle energy technique group. both of the groups have the conventional physical therapy in addition to these two interventions. data will be collect from the patients.30 minutes session twice a week will be given to the patients in each group. assessment will be done by using visual analog scale, Goniometer, Modified Oswestry Disability Index. Data will be entered and analyzed by using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* • Both genders

  * Between the ages group of 35-60 years
  * Patients with diagnosis of Sciatica.
  * Straight Leg Raise< 45°.
  * Having symptoms from past one month.

Exclusion Criteria:

* Inflammatory or other specific disorders of the spine such as ankylosing spondylitis, vertebral collapse, rheumatoid arthritis, stenosis, spondylolysthesis and osteoporosis.

  * History of any previous spinal surgical intervention
  * Symptomatic bilateral radiculopathy
  * Presence of any of red flags related to spinal column
  * History of involvement in any exercise program for lower extremity in recent time

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6 weeks
  For the assessment of pain, Visual Analogue Scale will be used. it is 0 to 10 cm where 0 means no pain 10 means sever pain
Goniometry | 6 weeks
  For the documentation of range of motion, straight leg raise test (SLR) will be used. For this purpose goniometer will use.
Modified Oswestry Disability Index | 6 weeks
  For the assessment of functional disability Modified Oswestry Disability Index will be used.

CONTACTS AND LOCATIONS:
Overall Officials: AHMAD Wassi, DPT, Principal Investigator — University of Lahore
Locations (1):
- Safi Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The IDP plane will be share with the researcher those are working on the same condition
Supporting Information: Study Protocol
Time Frame: Data sharing will b e available after the publication of the study
Access Criteria: Data assess will be provided via email to principal investigator Email:msptm02191002@student.uol.edu.pk

REFERENCES:
- See also: Effectiveness of surgery for sciatica with disc herniation is not substantially affected by differences in surgical incidences among three countries: results from the Danish, Swedish and Norwegian spine registries — http://link.springer.com/article/10.1007/s00586-018-5768-9
- See also: Characterization of the incidence and risk factors for the development of lumbar radiculopathy. Clinical Spine Surgery — http://onlinelibrary.wiley.com/doi/abs/10.1002/pri.1572